CLINICAL TRIAL: NCT03040661
Title: Randomized Trial of Femoral Vein Hemostasis After Ablation for Atrial Fibrillation With Manual Pressure Versus a Figure of 8 Suture
Brief Title: Femoral Vein Hemostasis After Ablation for Atrial Fibrillation With Manual Pressure Versus a Figure of 8 Suture
Acronym: Figure 8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-2381
Record Dates: First submitted 2017-01-24; First posted 2017-02-02 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Figure of 8 Suture (Experimental): Hemostasis after an ablation for atrial fibrillation with a figure of 8 suture.
  Interventions: Procedure: Ablation for atrial fibrillation.
- Manual Hemostasis Group (Active Comparator): Hemostasis after an ablation for atrial fibrillation with the Manual Hemostasis Technique.
  Interventions: Procedure: Ablation for atrial fibrillation.

INTERVENTIONS:
Procedure: Ablation for atrial fibrillation. — Ablation for atrial fibrillation.

SUMMARY:
Patients who undergo ablation for AF typically have 2 sheaths placed in each groin, including a large sheath when the Cryo Balloon is used for pulmonary vein isolation. During the procedure, heparin is administered to maintain a target ACT > 300 seconds. At the conclusion of the procedure, the venous sheaths are removed and hemostasis is obtained. There are at least 2 ways of obtaining hemostasis after venous access. In the manual hemostasis approach, an ACT is checked and protamine is administered. The ACT is rechecked 20" later, and if < 220 msec, the sheaths are pulled and hemostasis is achieved with manual pressure (Manual Hemostasis Group). Another approach is to place a Figure of 8 suture around the sheaths in each groin to achieve hemostasis as the sheaths are removed, and therefore obviate the need for assessment of the ACT, protamine administration, and manual pressure (Figure of 8 Group).

ELIGIBILITY:
Inclusion Criteria:

* Any patient who meets standard clinical criteria for an ablation of AF with Cryoballoon, and is to undergo the procedure

Exclusion Criteria:

1. Pregnant patients.
2. Age <18 years.
3. Patients who cannot provide consent in English.
4. Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Figure of 8 Suture | Manual Hemostasis Group
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Figure of 8 Suture | Manual Hemostasis Group | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.5) | 62.1 (9.4) | 62.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 21 | 22 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 30 | 31 | 61
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Time Required to Achieve Hemostasis
Description: Time Required to Achieve Hemostasis (minutes)
Time Frame: Time (minutes) from sheath removal till hemostasis achieved
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Figure of 8 Suture: Hemostasis after an ablation for atrial fibrillation with a figure of 8 suture.
  Ablation for atrial fibrillation.
- Manual Hemostasis Group: Hemostasis after an ablation for atrial fibrillation with the Manual Hemostasis Technique.
  Ablation for atrial fibrillation
Arm/Group | Figure of 8 Suture | Manual Hemostasis Group
Number analyzed (Participants) | 35 | 35
minutes | 0 (0) | 15 (6)

2. Primary Outcome: Time Required From the Completion of the Ablation Portion of the Procedure Until the Patient Leaves the EP Lab.
Description: Time required from the completion of the ablation portion of the procedure until the patient leaves the EP Lab (minutes)
Time Frame: Time (minutes) from completion of procedure till patient leaves room
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Figure of 8 Suture | Manual Hemostasis Group
Number analyzed (Participants) | 35 | 35
minutes | 20 (5) | 28 (9)

3. Secondary Outcome: Percent Groin Complications in Figure of 8 Suture Technique Group Compared to Manual Hemostasis Group
Description: Percent groin complications ( major or minor bleeding, additional pressure required for hemostasis, hematoma, pseudoaneurysm, and transfusion) in Figure of 8 suture technique group compared to manual hemostasis group.
Time Frame: Assessed after sheath removal till patient discharge
Measure: Number; unit: percent
Arm/Group | Figure of 8 Suture | Manual Hemostasis Group
Number analyzed (Participants) | 35 | 35
percent | 8.6 | 34.2

ADVERSE EVENTS:
Time Frame: In-hospital and 30 days post procedure
Arm/Group | Figure of 8 Suture | Manual Hemostasis Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 2/35 | 2/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Figure of 8 Suture (N=35) | Manual Hemostasis Group (N=35)
Hematoma or minor bleeding at site (Surgical and medical procedures) | 2 (35) | 2 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT03040661/Prot_SAP_000.pdf